CLINICAL TRIAL: NCT02577692
Title: Impact of Inspired Oxygen on Oxidative Stress and Breath Volatile Organic Compound Composition in Healthy Volunteers: A Randomized Controlled Cross-over Trial
Brief Title: Inspired Oxygen on Oxidative Stress and Breath Volatile Organic Compound Composition in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Klinikum der Universitaet Muenchen, Grosshadern (Other)
Collaborators: Airbus Defence and Space (Industry); DLR German Aerospace Center (Other)
Responsible Party: Principal Investigator, Michael Dolch, Dr. med., Klinikum der Universitaet Muenchen, Grosshadern
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: eN-2015-1.0
Record Dates: First submitted 2015-10-13; First posted 2015-10-16 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Oxidative Stress
MeSH Terms: interventions — Oxygen; Particulate Matter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen (Experimental): Day 1: breathing of 100% oxygen; Day 2: ambient air breathing
  Interventions: Other: Oxygen; Other: Ambient
- Ambient (Experimental): Day 1: breathing of 100% oxygen; Day 2: ambient air breathing
  Interventions: Other: Oxygen; Other: Ambient

INTERVENTIONS:
Other: Oxygen — breathing oxygen
Other: Ambient — breathing ambient air

SUMMARY:
High inspiratory oxygen fractions are known to induce oxidative stress and lipid peroxidation. The degrading products of oxidative stress induced lipid peroxidation are in part volatile and appear in breath where they can be measured non-invasively. However, there is lack of knowledge on the correlation of blood and breath biomarkers of oxidative stress.

This study aims to investigate the effects of a high inspiratory oxygen fraction on oxidative stress in healthy volunteers. The primary outcome is the appearance of exhaled breath biomarkers of oxidative stress by electrochemical sensors and ion mobility mass spectrometry. Secondary outcomes are changes in oxidative stress biomarkers in blood and their relationship to breath biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers who have given an oral and written informed consent

Exclusion Criteria:

* smoker or ex-smoker
* any pulmonary disease
* any heart disease
* any chemotherapy in the past
* any kind of daily medication

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Change in exhaled breath oxidative stress biomarker | 1, 4, and 24 hour
  Measurement of oxidative stress biomarkers in breath e.g. acetaldehyde, ethan, malondialdheyde, propionaldehyde, pentane

SECONDARY OUTCOMES:
Change in blood oxidative stress biomarkers | 1, 4, and 24 hour
  Measurement of oxidative stress biomarkers in blood e.g. ethane, malondialdehyde, pentane, propionaldheyde, total oxidative and antioxidative capacity, glutathione

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Dolch, MD, Principal Investigator — Klinikum der Universitaet Muenchen - Campus Grosshadern
Locations (1):
- Department of Aneshtesiology, University Hospital of Munich, München, Germany